CLINICAL TRIAL: NCT03961841
Title: A Randomised Controlled Trial Comparing Perioperative FLOT, FOLFOX and Preoperative Chemoradiation for Locally Advanced Esophagogastric Junction Adenocarcinoma
Brief Title: Perioperative Combination Chemotherapy Versus Chemoradiation for Locally Advanced EGJ Adenocarcinoma
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Sixth Affiliated Hospital, Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Jian Xiao, Deputy Director, Sixth Affiliated Hospital, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SAHMO202
Record Dates: First submitted 2019-05-22; First posted 2019-05-23 (Actual); Last update posted 2019-12-23 (Actual); Status verified 2019-12

CONDITIONS: Esophagogastric Junction Disorder; Neoplasms
MeSH Terms: conditions — Neoplasms | interventions — Chemoradiotherapy; Oxaliplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Chemoradiation (Active Comparator): weekly 5-Fu and oxaliplatin
  Interventions: Radiation: chemoradiation with weekly 5Fu and oxaliplatin
- FLOT (Experimental): Eight perioperative chemotherapy cycles
  Interventions: Drug: Perioperative mFLOT
- FOLFOX (Experimental): Twelve perioperative chemotherapy cycles
  Interventions: Drug: Perioperative FOLFOX

INTERVENTIONS:
Radiation: chemoradiation with weekly 5Fu and oxaliplatin — 5Fu 225 mg/m2 IV daily continuous infusion；oxaliplatin 40 mg/m2/week
  Arms: Chemoradiation
Drug: Perioperative mFLOT — Perioperative docetaxel 50mg/m2；oxaliplatin 85 mg/m2; 5Fu 2.4g/m2 civ 48 hours; repeated every 2 weeks; total of 8 cycles
  Arms: FLOT
Drug: Perioperative FOLFOX — Perioperative oxaliplatin 85 mg/m2; 5Fu 2.8g/m2 civ 48 hours; repeated every 2 weeks; total of 12 cycles
  Arms: FOLFOX

SUMMARY:
Patients with histologically confirmed esophagogastric junction adenocarcinoma with pre-operative staging cT3-4N+M0，aged between 18-75 years old, with adequate organ function and having an Eastern Cooperative Oncology Group performance status score ≤2, are randomized in a 1:1:1 ratio to receive neoadjuvant chemoradiotherapy with DT46-50Gy plus concomitant weekly oxaliplatin and 5-Fu, perioperative chemotherapy of FLOT regimen or FOLFOX regimen. The primary end point is disease free survival (DFS), and secondary end point is 5-year overall survival (OS), pathological complete remission (pCR) and treatment safety. The final study analytics are to be conducted at the end of the 5th year after the last patient's enrollment.

ELIGIBILITY:
Inclusion Criteria:

* informed consensus of the enrolled patients
* from 18 to 75 years old
* proven to be primary adenocarcinoma of EGJ
* pre-operative staging cT3-4N+M0
* no prior other chemotherapy and/or radiation against the disease
* normal function of all other vital organs including heart,liver ,kidney and so on
* Eastern Cooperative Oncology Group performance status: 0~2

Exclusion Criteria:

* history of other malignancy
* allergic reaction to capecitabine or oxaliplatin
* enrolled in other clinical trials
* abnormal GI tract function
* dysfunction of other organs
* pregnant or lactating females ,or refuse to receive contraception measures during chemotherapy
* other situations judged as not adaptive to the study by investigators

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 900 (Estimated)
Dates: Start 2020-06 (Estimated); Primary Completion 2024-08 (Estimated); Study Completion 2029-08 (Estimated)

PRIMARY OUTCOMES:
3 year of disease free survival | 3 year

SECONDARY OUTCOMES:
5 year of overall survival | 5 year
Rate of pathological complete remission | 1 year
Anastomosis leak rate | 1 year

IPD SHARING:
Plan to Share IPD: No